CLINICAL TRIAL: NCT02669381
Title: Dietary Phenylalanine Requirements During Different Stages of Gestation in Healthy Pregnant Women
Brief Title: Phenylalanine Requirements in Healthy Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H15-02558
Record Dates: First submitted 2015-11-30; First posted 2016-02-01 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Pregnancy
Keywords: Phenylalanine; Direct Amino Acid Oxidation; Stable isotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: phenylalanine intake (Other): Dietary supplement: phenylalanine intake
  Interventions: Dietary Supplement: Phenylalanine intake

INTERVENTIONS:
Dietary Supplement: Phenylalanine intake — Oral consumption of eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.

SUMMARY:
Phenylalanine is an essential amino acid that people need to obtain in their diets. Amino acids are the building blocks for protein, which is required to form tissues in the body. It is well known that pregnant women require more protein in their diets, but the exact amount for each amino acid is undetermined. To find out how much of phenylalanine pregnant women require, the investigators plan to study pregnant women in early and late gestation with a modern minimally invasive technique.

DETAILED DESCRIPTION:
The investigator's purpose is to determine the phenylalanine requirements in healthy pregnant women as part of a Master's Thesis project. The determined requirements can be taken into account when giving dietary recommendations, to ensure healthy pregnancies. The hypothesis is that the current recommendations for phenylalanine intake given to pregnant women are underestimated. The investigators also hypothesize that the phenylalanine requirements at early stages of pregnancy will be lower than the requirements towards the later stages of pregnancy.

Current dietary intake recommendations for phenylalanine are based on factorial (mathematical) calculations and do not account for requirement differences between early and late pregnancy. Static recommendations throughout all stages of pregnancy are not appropriate because of the multitude of adaptations the human body goes through during gestation. Whether phenylalanine requirements differ between different stages of gestation is unknown. In addition, phenylalanine is the precursor for tyrosine, which is a conditionally indispensable amino acid. Together they are referred to as the aromatic amino acids. The DRI gives a recommendation for total aromatic amino acids (TAA, phenylalanine + tyrosine) of 36 mg/kg/d during pregnancy. Since this study is the first interested in phenylalanine requirements during pregnancy, the investigators will determine the phenylalanine requirements in the presence of excess tyrosine (61 mg/kg/d) during pregnancy, similar to earlier studies.

The investigators will recruit healthy pregnant women aged 20 to 40 in their 13th-19th week of gestation or 33rd to 39th week of gestation. Once they get in contact with the lab, an initial visit (pre-study) will take place. Here, the participants will be measured for their eligibility and taken through the consent form. They have to participate in a pre-study for each stage of pregnancy, if they wish to participate in both stages. If they meet all the criteria and agree to participate, they will return for up to two study days per stage of 8 hours each. Therefore, if they are recruited during late pregnancy they are only able to participate in two study days in total. During these study days they will be fed protein shakes containing the stable isotope, and then oxidation of this isotope will be measured to determine a breakpoint (requirement) of phenylalanine. Breath samples, urine samples, and a small blood sample will be taken during the study day.

ELIGIBILITY:
Inclusion Criteria:

* over the age of twenty
* under the age of forty
* in overall good health
* pregnant with a single child

Exclusion Criteria:

* Be under the age of twenty
* Be over the age of forty
* Be pregnant with more than one child
* Have a history of cardiovascular disease, endocrine disorders, or metabolic disorders
* Have recently lost a substantial amount of weight
* Delivered a baby in the last 18 months
* Be substance dependent
* Be allergic to eggs
* Have severe nausea through the pregnancy
* Have gestational diabetes
* Have a history of spontaneous abortions
* Have had an unhealthy pre-pregnancy body mass index

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
13C Phenylalanine Oxidation | 8 hours
  Urine, breath and a single blood sample will be collected during the study to measure the rate of oxidation of 13C phenylalanine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, Ph.D., Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ennis MA, Rasmussen BF, Lim K, Ball RO, Pencharz PB, Courtney-Martin G, Elango R. Dietary phenylalanine requirements during early and late gestation in healthy pregnant women. Am J Clin Nutr. 2020 Feb 1;111(2):351-359. doi: 10.1093/ajcn/nqz288. PMID 31758682